CLINICAL TRIAL: NCT00004101
Title: Phase I Trial of Humanized 1D10 Monoclonal Antibody (Hu1D10) In Patients With Relapsed Non-Hodgkin's Lymphoma (NHL)
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Recurrent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067318; UIHC-UICC-LW-02; NCI-T99-0019
Record Dates: First submitted 1999-12-10; First posted 2004-05-03 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2001-05

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — apolizumab

ARMS (1):
- Arm I (Experimental): Patients receive monoclonal antibody Hu1D10 IV over 2-4 hours on days 1, 8, 15, and 22. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of monoclonal antibody Hu1D10 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 6 patients experience dose limiting toxicity. Once the MTD is determined, an additional cohort of 3-6 patients receive Hu1D10 IV over 2-4 hours on days 1-5.
  Interventions: Biological: apolizumab

INTERVENTIONS:
Biological: apolizumab

SUMMARY:
Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have recurrent non-Hodgkin's lymphoma. Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Assess the safety and tolerability of monoclonal antibody Hu1D10 in patients with previously treated non-Hodgkin's lymphoma expressing the antigen recognized by Hu1D10.

II. Determine the maximum tolerated dose of monoclonal antibody Hu1D10 in these patients.

III. Evaluate the pharmacokinetics, compare the pharmacology at different dose levels, and determine the optimal biological dose of this drug in these patients.

IV. Evaluate any antilymphoma effects of this drug in these patients.

OUTLINE: This is a dose escalation, multicenter study.

Patients receive monoclonal antibody Hu1D10 IV over 2-4 hours on days 1, 8, 15, and 22. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of monoclonal antibody Hu1D10 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 6 patients experience dose limiting toxicity. Once the MTD is determined, an additional cohort of 3-6 patients receive Hu1D10 IV over 2-4 hours on days 1-5.

Patients are followed at 4 weeks, 50 days, and periodically thereafter until disease progression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-Hodgkin's lymphoma in relapse or refractory to prior treatment
* At least 50% of malignant cells on biopsy specimen reactive with the 1D10 antibody OR at least 50% of B cells within tumor reactive with 1D10 if extensive T cell infiltrations present
* Measurable or evaluable disease
* Circulating tumor cells fewer than 5,000/mm3 (in dose escalation phase only)
* Not eligible for curative conventional therapy

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0-2
* Life expectancy: At least 3 months
* Platelet count at least 75,000/mm3
* Bilirubin less than 2.5 mg/dL
* SGOT less than 3 times upper limit of normal
* Creatinine less than 2.0 mg/dL
* No New York Heart Association class III or IV heart disease
* No clinically significant pulmonary disease
* No active serious infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception HIV negative

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior interferon
* Concurrent transfusions allowed
* At least 4 weeks since prior cytotoxic chemotherapy
* No concurrent antineoplastic agents
* At least 4 weeks since prior corticosteroids
* No concurrent glucocorticoids
* At least 4 weeks since prior radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 1999-11; Primary Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Link, MD, Study Chair — Holden Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Biologics Evaluation Section, Bethesda, Maryland
  - New York Presbyterian Hospital - Cornell Campus, New York, New York

REFERENCES:
- [Result] Link BK, Wang H, Byrd JC, et al.: Phase I trial of humanized 1D10 (Hu1D10) monoclonal anitbody class II molecules in patients with relapsed lymphoma. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A86, 2000.